CLINICAL TRIAL: NCT04306731
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Assess the Use of Nanotechnology Structured Water Magnalife for the Prevention of Recurrent Urinary Tract Infections.
Brief Title: Effect of Nanotechnology Structured Water Magnalife for the Prevention of Recurrent Urinary Tract Infections.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, ALI KAMAL M. SAMI, Principal investigator, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: College of Medicine
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: nanotechnology water, antibiotic prophylaxis, recurrent UTI.
MeSH Terms: conditions — Urinary Tract Infections | interventions — Trimethoprim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional (Group M) (Experimental): The group of patients given nanotechnology structured water magnalife
  Interventions: Dietary Supplement: Nanotechnology Structured water Magnalife
- Control (Group T) (Active Comparator): The group of patients given Trimethoprim
  Interventions: Drug: Trimethoprim
- Placebo (Group O) (Placebo Comparator): The group of patients given ordinary bottled drinking water
  Interventions: Dietary Supplement: Ordinary bottled drinking water

INTERVENTIONS:
Dietary Supplement: Nanotechnology Structured water Magnalife — Nanotechnology Structured water Magnalife is drinking water that has been modified using nanotechnology to change the structuring of water molecules
  Other Names: Magnalife; 5200250040466
  Arms: Interventional (Group M)
Drug: Trimethoprim — Antibiotic
  Other Names: Proloprim
  Arms: Control (Group T)
Dietary Supplement: Ordinary bottled drinking water — Placebo
  Arms: Placebo (Group O)

SUMMARY:
This study investigates nanotechnology structured water magnalife in urology and to test its effects against lower urinary tract infections (UTI) in females.

DETAILED DESCRIPTION:
This study represents the first time to use nanotechnology structured water magnalife in urology and to test its effects against lower urinary tract infections (UTI) in females. Urinary tract infection (UTI ) is the second most common bacterial infection, affecting women at a much higher frequency than men. There is a higher rate of recurrence of UTI, and a recurrent infection will follow 25-35% of initial UTI episodes within 3-6 months.

Intermittent or prolonged low dose antibiotic therapy has been used to treat and prevent recurrent UTI. Emerging of resistance to antimicrobial agents, enormous economic burden, and the side effects of antibiotics have led to the search for an alternative non-antibiotic prophylaxis of recurrent UTI. Nanotechnology structured water is a new type of drinking water that has been prepared using different types of energy fields and electromagnetic fields to produce this structured water, which has new and different characteristics from the ordinary water.

In the current study, the efficacy of nanotechnology structured water magnalife was compared with low-dose Trimethoprim and bottled drinking water for the prevention of recurrent UTI.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 2 (two or more than two) UTI in the last 6 months
* ≥ 3 (three or more than three) UTI in the last 12 months

Exclusion Criteria:

* immunotherapy
* radiotherapy
* malignancy
* steroids
* chronic infections
* chemotherapy
* immunosuppressive drugs
* anatomical abnormality of the urinary tract
* surgical operation the urinary tract

Ages: 24 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2014-09-20 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
Recurrent Urinary Tract Infection | Twelve months
  Urinalysis by GUE (>10 white blood cells (WBC)/mm3 per high-power field (HPF) Urine culture (urinary pathogen of ≥105 colony-forming units (CFU) per mL)

SECONDARY OUTCOMES:
Time to first recurrent UTI | Twelve months
  The time since the beginning of the study until the first recurrent UTI (days)

CONTACTS AND LOCATIONS:
Overall Officials: Ali K M.Sami, Ph.D., Principal Investigator — College of Medicine, University of Sulaimani
Locations (1):
- College of Medicine, University of Sulaimani, Sulaymaniyah, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No
The duration of illness, number of recurrence of UTI, other co-morbid diseases